CLINICAL TRIAL: NCT06611774
Title: Metabolic Syndrome in Patients with Knee Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady kerollos louis shamroukh, assistant lecturer, Assiut University
Other Study IDs: osteoarthritis MetSyndrome
Record Dates: First submitted 2024-08-09; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Metabolic Syndrome
Keywords: knee osteoarthritis; metabolic syndrome
MeSH Terms: conditions — Osteoarthritis, Knee; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Study the prevalence of metabolic syndrome in patients with knee osteoarthritis and conclude the relationship between metabolic syndrome and the severity of knee osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis is one of the most common clinical conditions causing severe chronic and restrictive disability, especially in elderly people.

Of those aged 60 years and older, 10% of men and 13% of women had symptomatic knee OA . As the population ages and the prevalence of obesity and overweight generaly rises , the percentage of persons affected with symptomatic knee OA will likely increase.

The clinical manifestations in patients are joint pain, stiffness, and functional limitation .

Among all body joints; knee joint is the most commonly affected joint with osteoarthritis and accounts almost for four-fifth of the osteoarthritis burden worldwide .

Epidemiological research has shown an encouraging relationship between OA and metabolic syndrome , MetS include hypertension, dyslipidemia, hyperglycemia, and obesity .Recently, metabolic OA has been nominated as the fifth component of MetS .

Studies reported that adipokines may contribute to the development of osteoarthritis (OA) by increasing inflammatory cytokines and growth factors, modifying insulin sensitivity, and triggering processes that break down cartilage.

Studies also reported that hypertension can be linked to osteoarthritis through astherosclerosis which cause subchondral bone ischemia accelerating OA progression.

Furthermore, researches have linked glucose levels to knee osteoarthritis , supporting the possibility of pathophysiological mechanisms such oxidative stress in the chondrocytes and Cartilage-associated production of advanced glycation end products (AGEs) .

ELIGIBILITY:
Inclusion

1. Both males and female .
2. Age between 30 and 70 years old.
3. Patient fulfill the criteria of knee osteoarthritis .

Exclusion Criteria:

1. Patients known to have rheumatological disease .
2. Patients with meniscal or cruciate ligament injury .
3. Patients with previous knee surgery .

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in assiut university hospitals and presenting to its clinics
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome in patients with knee osteoarthritis | Baseline
  Study the prevalence of metabolic syndrome in patients with knee osteoarthritis and the relation between metabolic syndrome and clinical, functional, radiological finding of knee osteoarthritis

REFERENCES:
- [Background] Maddah S, Mahdizadeh J. Association of Metabolic Syndrome and Its Components with Knee Osteoarthritis. Acta Med Iran. 2015 Dec;53(12):743-8. PMID 26749230
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Goldring SR, Goldring MB. Changes in the osteochondral unit during osteoarthritis: structure, function and cartilage-bone crosstalk. Nat Rev Rheumatol. 2016 Nov;12(11):632-644. doi: 10.1038/nrrheum.2016.148. Epub 2016 Sep 22. PMID 27652499
- [Background] Xie DX, Wei J, Zeng C, Yang T, Li H, Wang YL, Long HZ, Wu ZY, Qian YX, Li KH, Lei GH. Association between metabolic syndrome and knee osteoarthritis: a cross-sectional study. BMC Musculoskelet Disord. 2017 Dec 16;18(1):533. doi: 10.1186/s12891-017-1890-9. PMID 29246142
- [Background] Courties A, Sellam J. Osteoarthritis and type 2 diabetes mellitus: What are the links? Diabetes Res Clin Pract. 2016 Dec;122:198-206. doi: 10.1016/j.diabres.2016.10.021. Epub 2016 Nov 5. PMID 27889689
- [Background] Tu C, He J, Wu B, Wang W, Li Z. An extensive review regarding the adipokines in the pathogenesis and progression of osteoarthritis. Cytokine. 2019 Jan;113:1-12. doi: 10.1016/j.cyto.2018.06.019. Epub 2018 Jun 28. PMID 30539776